CLINICAL TRIAL: NCT06598514
Title: Effect of Chlorhexidine Perineal Lavage Following Defecation in Post-Menopausal Women With Recurrent Urinary Tract Infection
Brief Title: Chlorhexidine Lavage for Recurrent Urinary Tract Infection
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sara Cichowski, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00027352
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Urinary Tract Infections; Recurrent Urinary Tract Infection
Keywords: Menopause
MeSH Terms: conditions — Urinary Tract Infections | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Individuals meeting inclusion criteria will be randomized to the treatment (2% chlorhexidine perineal lavage following defecation) or control (sterile water perineal lavage following defecation) and rates of urinary tract infection will be compared. Balanced randomization will be performed via computer-generated assignments in REDCap with random permuted blocks varying in size between 8 and 10.
Who Masked: Participant
Masking Description: Participants will be blinded to their assigned treatment. All participants will receive a box containing their randomized intervention and identical use instructions. Opaque bottles will contain either a sterile water solution or 2% chlorhexidine. Spray bottles will be identical in external appearance.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine Lavage (Experimental): 2% chlorhexidine perineal lavage following defecation
  Interventions: Drug: Chlorhexidine
- Sterile Water Lavage (Active Comparator): Sterile water perineal lavage following defecation
  Interventions: Drug: Sterile Water

INTERVENTIONS:
Drug: Chlorhexidine — Participants will use a 2% chlorhexidine perineal lavage following defecation
  Arms: Chlorhexidine Lavage
Drug: Sterile Water — Participants will use a sterile water perineal lavage following defecation
  Arms: Sterile Water Lavage

SUMMARY:
A two-arm randomized control trial evaluating rates of urinary tract infection in post-menopausal women on vaginal estrogen with recurrent urinary tract infections.

DETAILED DESCRIPTION:
There is a critical need for low-cost, non-antibiotic interventions that are feasible for patients to utilize for risk reduction and prevention of recurrent urinary tract infections (UTIs). The current most effective non-antibiotic prophylaxis for recurrent UTI is vaginal estrogen; however, approximately 50% of women will continue to experience UTIs. The investigators propose a randomized control trial of postmenopausal women on vaginal estrogen with the diagnosis of recurrent UTIs to evaluate a novel post-defecation hygienic strategy utilizing a 2% chlorhexidine perineal lavage. Participants will be randomized to either a 2% chlorhexidine perineal lavage or a water lavage. Study participants will be followed for up to 6-months, and UTIs will be tracked with culture proven samples throughout study participation.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female between age 55 and 89
* No post-menopausal bleeding
* Diagnosis of recurrent urinary tract infection (UTI) in the electronic health record or as two culture proven UTIs in 6 months or three culture proven UTIs in 12 months
* At least one UTI in the 6 months prior to entering the study
* Asymptomatic for UTI symptoms at the time of enrollment.
* On vaginal estrogen therapy for at least 6 weeks prior to enrollment
* Ready access to email and internet

Exclusion Criteria:

* Recent prophylactic antibiotic use (washout period of 4 weeks)
* Neurogenic bladder
* Diagnosis of urinary retention
* Uncorrected Stage III-IV prolapse
* Indwelling catheter or need for intermittent self-catheterization
* History of complicated UTIs
* History of interstitial cystitis or bladder pain syndrome
* History of fecal incontinence/accidental bowel leakage
* Greater than 14 bowel movements per week
* Non-English speaking
* Allergy to chlorhexidine gluconate
* Inability to utilize vaginal estrogen therapy
* Recent urogynecological or urologic surgery (<12 weeks)

Ages: 55 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Urinary Tract Infection (UTI) | 90 days following treatment initiation
  The proportion of participants in each arm who experience a urinary tract infection (UTI) within 90 days will be compared

SECONDARY OUTCOMES:
Vulvovaginal Symptom Questionnaire (VSQ) | VSQ administered prior to randomization and at 6 weeks, 12 weeks, and 24 weeks post-randomization
  Vulvovaginal symptoms will be evaluated using the VSQ from baseline to post-intervention and compared between the groups with and without chlorhexidine in their perineal lavage. The VSQ is scored on a scale of 0-16 for those who are not sexually active or 0-20 for those who are sexually active, with a higher score indicating worse outcomes.
Urinary Distress Inventory (UDI-6) | UDI-6 administered prior to randomization and at 6 weeks, 12 weeks, and 24 weeks post-randomization
  Urinary symptoms will be evaluated using the UDI-6 from baseline to post-intervention and compared between the groups with and without chlorhexidine in their perineal lavage. It is scored on a scale from 0 to 100 with higher scores indicating worse outcomes.

OTHER OUTCOMES:
Participant Satisfaction with Virtual Recruitment | Upon completion of the intervention period, 90 days after randomization
  Satisfaction with virtual recruitment and enrollment will be evaluated using the Patient Global Impression scales to allow for participant reported outcomes regarding perceived change following intervention. It is scored on a scale from 1 to 7 with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States